CLINICAL TRIAL: NCT02002000
Title: Chronic Pain and Vitamin D: a Randomized Pilot Study in General Practice
Brief Title: Chronic Pain and Vitamin D
Acronym: DOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-802
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Musculoskeletal Pain; Vitamin D Supplementation
Keywords: Vitamin D deficiency; Musculoskeletal pain; Vitamin D supplementation
MeSH Terms: conditions — Vitamin D Deficiency; Musculoskeletal Pain | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Experimental): Patients receiving 3 doses of vitamin D (cholecalciferol)
  Interventions: Drug: vitamin D (cholecalciferol)
- Placebo (Experimental): Patients receiving 3 doses of placebo according to the same schedule as experimental arm
  Interventions: Drug: Placebo, similar in appearance and taste to cholecalciferol

INTERVENTIONS:
Drug: vitamin D (cholecalciferol) — Patients from the vitamin D arm will receive an orally supplementation of 600 000 UI cholecalciferol in 3 doses: 200 000 UI at baseline (day 1), 200 000 UI on day 15 and 200 000 UI on day 30. Cholecalciferol will be presented in blisters, in a non-differentiable form in appearance and taste from placebo, either for the patient or the doctor
  Arms: vitamin D
Drug: Placebo, similar in appearance and taste to cholecalciferol — Patients from the placebo arm will receive 3 doses of placebo to be taken orally: one at baseline (day 1), one on day 15, one on day 30. Placebo will be presented in blisters in a non-differentiable form in appearance and taste from cholecalciferol either for the patient or the doctor.
  Arms: Placebo

SUMMARY:
Non-systematized chronic musculoskeletal pains are a frequent reason for consulting in general practice. The possible causes are numerous and sometimes nonspecific. In some cases, the etiologic investigation of patients with non-systematized and chronic musculoskeletal pain can not highlight any organic cause. Several studies have shown a link between these symptoms and vitamin D deficiency, characterized by a blood level of 25 (OH) vitamin D < 20.8ng/ml. This deficit is easy to identify and to correct through proper vitamin D supplementation with few side effects. Nevertheless, it remains unknown and vitamin D deficiency is rarely considered as a possible etiology in patients with chronic pain. We hypothesize that vitamin D supplementation in patients with non-systematized musculoskeletal pain and deficient in vitamin D could improve painful symptoms. We aim to perform a double-blind randomized controlled trial, vitamin D versus placebo, to assess the pain improvement after vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* Aged 18-50 years (included)
* Consulting their general practitioner
* With chronic and diffuse musculoskeletal pain, without known etiology, lasting for at least 3 months
* With a 25(OH)vitamin D deficiency <20.8 ng/ml (52 nmol/l) at inclusion
* Who signed the consent form

Exclusion Criteria:

* Identifiable source of pain requiring an appropriate specific management
* Disease or treatment that may interfere with the metabolism of vitamin D
* Current or previous hypercalcemia or hypercalciuria, treatment with digitalics and patients with history of nephrolithiasis
* Current treatment with vitamin D or at least one vitamin D vial taken over the previous 6 months
* Pregnancy or breastfeeding
* not affiliated to a social security system
* Refusal or inability to give consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in the two groups who reported a decrease in the overall pain after 3 months of treatment with vitamin D versus placebo. | 3 months after inclusion
  item 5 of the Brief Pain Inventory will be measured in each patient to assess the overall pain score at inclusion and after 3 month of treatment with vitamin D or placebo

SECONDARY OUTCOMES:
: Proportion of patients in both groups reporting an evolution of the minimum and the maximum of intensity of pain | 3 months after inclusion
  item 3 and 4 of the Brief Pain Inventory will be measured in each patient to assess the minimum and the maximum pain scores at inclusion, after 45 days and after 3 months of treatment with vitamin D or placebo
Proportion of patients in both groups reporting a decrease in the impact of pain on daily activities | 3 months after inclusion
  item 9 of the Brief Pain Inventory will be measured in each patient to assess the score of the impact of pain on daily activities at inclusion, after 45 days and after 3 months of treatment with vitamin D or placebo
Proportion of patients reporting a decrease in the consumption of analgesic drugs | 3 months after inclusion
  Patients of both groups will be asked at inclusion, after 45 days and after 3 months, if they took analgesic drugs: name, class and dose of each treatment will be registered in a standardized questionnaire
Proportion of patients in both groups reporting a decrease in the consumption of care (consultations and work stoppages) | 3 months after inclusion
  Patients of both groups will be asked at inclusion, after 45 days and after 3 months, if they consulted any health care professional : which health care professional, how many time, the reason for consultation and work stoppages will be registered in a standardized questionnaire
Proportion of patients in both groups reporting an improvement in quality of life | 3 months after inclusion
  Quality of life will be measured in patients of both groups by the SF-36 questionnaire, at inclusion and after 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie SCHOTT, Pr, Principal Investigator — Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon
Locations (1):
- Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon, Lyon, France